CLINICAL TRIAL: NCT03115385
Title: Probiotics and the Gut Microbiome in Obese Hispanic Youth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funds ended.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael I. Goran, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HS-14-00683
Record Dates: First submitted 2017-03-29; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Obesity, Abdominal; Adiposity
MeSH Terms: conditions — Obesity, Abdominal; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Inactive ingredients include maltose, lemon flavoring (or corn starch if unflavored), and silicon dioxide.
  Interventions: Dietary Supplement: Placebo
- VSL#3 (Active Comparator): VSL#3 is classified as a medical food that is specially formulated and processed to provide a precise mixture of 8 strains of bacterial species with potential synergistic relationships. These strains include Streptococcus thermophilus, Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, and Lactobacillus delbrueckii subsp. bulgaricus.
  Interventions: Dietary Supplement: VSL#3

INTERVENTIONS:
Dietary Supplement: VSL#3 — VSL#3 will provide active packets. Subjects will take 2 to 3 packets per day with for 16 weeks. The study team will supply each participant with all necessary packets on a weekly or bi-weekly basis within 1-2 weeks after their first visit. VSL#3 probiotic is provided in powder form and needs to be mixed with cold, non-fizzy liquid for consumption. For this reason, the study team will also provide participants with zero calorie sugar fee beverages to mix their packet with (e.g., vitamin water zero with stevia).
  Arms: VSL#3
Dietary Supplement: Placebo — A matched placebo to VSL#3 will be provided. The placebo will be identical to the active VSL#3 probiotic in aspects such as packaging, color, taste, texture, shape, and odor. The placebo will not contain active ingredients. The study team will supply each participant with all necessary packets on a weekly or bi-weekly basis within 1-2 weeks after their first visit. The placebo is provided in powder form and needs to be mixed with liquid for consumption. For this reason, the study team will also provide participants with zero calorie sugar fee beverages to mix their packet with (e.g., vitamin water zero).
  Arms: Placebo

SUMMARY:
This study will recruit 40 obese Hispanic youth (12 - 18 years of age who are greater than or equal to Tanner stage 4) from hospitals, clinics, and community centers. Participants will be randomly assigned to 16 weeks of probiotics (3 packets/day of VSL#3) or matched placebo. The purpose of this study is to demonstrate through a proof-of-concept trial that probiotics have the potential to alter the gut microbiome and gut hormones.

DETAILED DESCRIPTION:
Recent studies suggest that probiotic supplementation has the potential to restore gut microbiota homeostasis and reduce fatty liver. No studies have examined the effects of probiotic supplementation on the gut microbiome in obese Hispanic youth who are increased risk of type 2 diabetes and fatty liver. Therefore, the investigator proposes a double-blind randomized trial of probiotic supplementation in obese Hispanic youth in order to determine if probiotic supplementation results in alterations to the gut micro biome. The purpose of this study is to demonstrate through a proof-of-concept trial that probiotics have the potential to alter the gut microbiome and gut hormones. As a secondary aim the investigator will examine wether any changes in the gut microbiome are related to changes in liver fat, fibrosis, glycemia, or body weight. The study team will recruit 40 obese Hispanic youth (12 - 18 years of age who are greater than or equal to Tanner stage 4) from hospitals, clinics, and community centers. The studies primary outcome is alterations in the composition of the gut microbiome which will be examined through fecal and blood bacterial profiling (16S DNA targeted metagenomics), markers of gut permeability/bacterial translocation, and gut derived hormones involved with appetite regulation (GLP-1, peptide YY, ghrelin). Secondary outcomes include liver fat and liver fibrosis (MR elastography), total body fat (DEXA), visceral fat (MRI). Participants will be randomly assigned to 16 weeks of probiotics (3 packets/day of VSL#3) or matched placebo. The main effects of the intervention will be evaluated in a general linear model, with change in outcomes as the dependent variable and active intervention group as the independent variable. Covariates will include sex, BMI percentile, the baseline value of the outcome variable, as well as baseline factors found to differ among groups. Post hoc pairwise comparisons of the two groups will adjust for multiple comparisons using a Tukey correction.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Obese (BMI percentile ≥95th for age and gender)
* Hispanic males and females who are 12-18 years of age and are ≥Tanner Stage 4.

Exclusion Criteria:

Participants will be excluded from the study if any of the following apply:

1. diagnosis of any disease that is known to influence insulin action and secretion (including type 1 and 2 diabetes);
2. current or past involvement in any weight loss, exercise, or sports program in the six months prior to participation
3. use of medication known to influence body composition or fat distribution (e.g. Cushing syndrome), insulin resistance, gut function, or lipid profiles;
4. history of renal / liver disease or any disease affecting liver fibrosis and steatosis;
5. diagnosis/current treatment for celiac, inflammatory bowel disease, Crohn's disease or other major GI issues;
6. those who are immune compromised;
7. pregnancy;
8. current smoking (more than 1 cigarette in the past week), >200 cigarettes in lifetime, or use of other recreational drugs;
9. alcohol consumption;
10. other siblings in the study;
11. physician diagnosis of major illness or eating disorder;
12. physical/cognitive handicaps preventing participation;
13. and recent antibiotic treatment (within the previous 30 days).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2015-05-30 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

PRIMARY OUTCOMES:
Change in abundance of gut microbiome and gut hormones measured pre and post blood and stool sample collections. | 16 weeks
  To determine whether probiotic (VSL#3) supplementation affects gut microbiome and gut hormones involved with appetite regulation in obese young Hispanics.

SECONDARY OUTCOMES:
Interaction between gut microbiome and liver fat, fibrosis, obesity, and glycemia measured pre and post blood and stool sample collections and through Dxa and MRI scans.. | 16 weeks
  To determine whether there are any relationships between changes in the gut microbiome and changes in liver fat, fibrosis, obesity, and glycemia after 16 weeks of probiotic supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang B, Sang L, Wang Y, Tong J, Zhang D, Wang B. The protective effect of VSL#3 on intestinal permeability in a rat model of alcoholic intestinal injury. BMC Gastroenterol. 2013 Oct 20;13:151. doi: 10.1186/1471-230X-13-151. PMID 24138544
- [Result] Alisi A, Bedogni G, Baviera G, Giorgio V, Porro E, Paris C, Giammaria P, Reali L, Anania F, Nobili V. Randomised clinical trial: The beneficial effects of VSL#3 in obese children with non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2014 Jun;39(11):1276-85. doi: 10.1111/apt.12758. Epub 2014 Apr 16. PMID 24738701
- [Result] Eslamparast T, Eghtesad S, Hekmatdoost A, Poustchi H. Probiotics and Nonalcoholic Fatty liver Disease. Middle East J Dig Dis. 2013 Jul;5(3):129-36. PMID 24829682
- [Result] Rajkumar H, Mahmood N, Kumar M, Varikuti SR, Challa HR, Myakala SP. Effect of probiotic (VSL#3) and omega-3 on lipid profile, insulin sensitivity, inflammatory markers, and gut colonization in overweight adults: a randomized, controlled trial. Mediators Inflamm. 2014;2014:348959. doi: 10.1155/2014/348959. Epub 2014 Mar 26. PMID 24795503
- [Result] Delzenne NM, Neyrinck AM, Backhed F, Cani PD. Targeting gut microbiota in obesity: effects of prebiotics and probiotics. Nat Rev Endocrinol. 2011 Aug 9;7(11):639-46. doi: 10.1038/nrendo.2011.126. PMID 21826100
- [Result] Wong VW, Won GL, Chim AM, Chu WC, Yeung DK, Li KC, Chan HL. Treatment of nonalcoholic steatohepatitis with probiotics. A proof-of-concept study. Ann Hepatol. 2013 Mar-Apr;12(2):256-62. PMID 23396737
- [Result] Kootte RS, Vrieze A, Holleman F, Dallinga-Thie GM, Zoetendal EG, de Vos WM, Groen AK, Hoekstra JB, Stroes ES, Nieuwdorp M. The therapeutic potential of manipulating gut microbiota in obesity and type 2 diabetes mellitus. Diabetes Obes Metab. 2012 Feb;14(2):112-20. doi: 10.1111/j.1463-1326.2011.01483.x. Epub 2011 Nov 22. PMID 21812894
- [Result] Wang J, Tang H, Zhang C, Zhao Y, Derrien M, Rocher E, van-Hylckama Vlieg JE, Strissel K, Zhao L, Obin M, Shen J. Modulation of gut microbiota during probiotic-mediated attenuation of metabolic syndrome in high fat diet-fed mice. ISME J. 2015 Jan;9(1):1-15. doi: 10.1038/ismej.2014.99. Epub 2014 Jun 17. PMID 24936764